CLINICAL TRIAL: NCT05626725
Title: An Observational Study to Assess the Safety and Effectiveness of Automated Insulin Delivery (AID) Systems in Physically Active Adults with Type 1 Diabetes in Free-living Conditions (AIDE-1)
Brief Title: Safety and Effectiveness of Automated Insulin Delivery (AID) Systems in Physically Active Adults with Type 1 Diabetes
Acronym: AIDE-1
Status: Recruiting | Type: Observational
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, MD, PhD, PROMD platform director, Clinic VP, Institut de Recherches Cliniques de Montreal
Other Study IDs: 2023-1190
Record Dates: First submitted 2022-09-09; First posted 2022-11-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observationnal cohort: Patients with type 1 diabetes and using an AID system.
  Interventions: Device: Automated insulin delivery system

INTERVENTIONS:
Device: Automated insulin delivery system — This is an outpatient prospective observational study to evaluate the effect of DIY-AID use on maintaining glucose levels in physically active adult people living with T1D.

SUMMARY:
Despite recent medical and technological advances, optimal glycemic control (time in range; TIR) and prevention of hypoglycemia remain significant challenges for people living with type 1 diabetes (T1DM). Automated insulin delivery systems (AIDs) combine an insulin pump coupled via an algorithm with a continuous glucose monitor (CGM), allowing constant adjustment of insulin doses according to blood glucose levels. Despite the significant improvement in blood glucose parameters and quality of life with these systems, they are not available to everyone and more and more people with diabetes are resorting to home-made or do-it-yourself (DIY) systems to access this technology. DIY systems are not approved or regulated by Health Canada, despite the growing interest. There have been no studies looking at this type of system in active people living with DbT1, including the risk of exercise-induced hypoglycemia.

The primary objective of this study is to evaluate the safety and efficacy of IDA systems in physically active individuals living with type 1 diabetes.This is a real-life observational study in people with commercial IDA (control group) and IDA-DIY. This study includes only one inclusion visit (which may be virtual) and the observation period is 6 weeks.

Participants will be required to wear their own artificial pancreas system and give us access to blood glucose and insulin data at the end of the study. They will be required to wear a watch to record physical activity (FitBit). We will ask them to complete information about their diet at least twice a week for a whole day (Keenoa application).

Finally, participants will be asked to complete a physical activity diary to complete data (carbohydrates in prevention of activity, insulin suspension, hypoglycemia during or after exercise, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥ 18 years old.
2. Clinical diagnosis of type 1 diabetes or latent autoimmune diabetes in adults (LADA) for at least one year. (The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.)
3. Using automated insulin delivery systems (Commercial or DIY) for at least 3 months.
4. Willing to share CGM data and insulin pump data with the research team. This access will be limited to the study period.
5. Exercising at least twice weekly (Questionnaire assessment MAQ) or willing to exercise at least twice weekly during the study period.
6. Willing to share physical activity tracker data with the research team and if applicable, data about the menstrual cycle.

Exclusion Criteria:

1. Do not understand French or English
2. Anticipated therapeutic change (including change of insulin type [switching to biosimilar is acceptable] and/or type of CGM sensor) between admission and end of the study.
3. Anticipated need to use acetaminophen (dose above 1g every 6 hours) or vitamin C (dose above 500mg DIE) between admission and end of the study.
4. Pregnancy (ongoing or current attempt to become pregnant).
5. Breastfeeding.
6. Uncontrolled thyroid disease (recent less than 5 months TSH should be in target range and treatment stable for at least 6 weeks).
7. Severe hypoglycemic episode within two weeks of screening.
8. Severe hyperglycemic episodes requiring hospitalization in the last 3 months
9. Current use of glucocorticoid medication (except low stable dose and inhaled steroids and stable adrenal insufficiency treatment e.g., Cortef®).
10. Current use of adjunct therapy such as SGLT-2 inhibitors or GLP_1 receptor analog unless at a stable dose for at least 3 months, without anticipated change during the study and appropriate ketone testing is performed in case of off-label SGLT2 usage.
11. Anticipated radiologic examination incompatible with CGM wear for more than 10 days between admission and end of the study (e.g., repeated MRI).
12. Physically inactive participants (see inclusion criteria #5).
13. People with professional activities involving night shifts, as it may influence glycemic profiles differently compared to people working days and sleeping nights.
14. In the opinion of the investigator, a participant who is unable or unwilling to complete the study (e.g., recent injury, foot wound, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes using an AID system; Physically active
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose levels from start of exercise to nadir during or up to 30 min post exercise. | 6 weeks
  nadir: the lowest point on a glucose curve

SECONDARY OUTCOMES:
Hypoglycemic events (n) 120-min before, during and 120-min after recorded structured PA sessions | 6 weeks
  Number of hypoglycemic events
Hypoglycemic events (n) during (at least 15-min) of habitual PA and 30-min after | 6 weeks
  Number of hypoglycemic events
Time in range 120-min before, during and 120-min after recorded structured PA sessions | 6 weeks
  Time (min and percentage) with glucose levels a. between 3.9 and 10.0 mmol/L; b. below 3.9 mmol/L; c. below 3.0 mmol/L; d. above 10.0 mmol/L
Time in range during (at least 15-min) of habitual PA and 30-min after | 6 weeks
  Time (min and percentage) with glucose levels a. between 3.9 and 10.0 mmol/L; b. below 3.9 mmol/L; c. below 3.0 mmol/L; d. above 10.0 mmol/L
CHO intake 120-min before, during and 120-min after recorded structured PA sessions | 6 weeks
  Carbohydrate intake (g), timing and purpose of CHO intake prior to, during and within 30-min following PA.mmol/L; b. below 3.9 mmol/L; c. below 3.0 mmol/L; d. above 10.0 mmol/L
CHO intake during (at least 15-min) of habitual PA and 30-min after | 6 weeks
  Carbohydrate intake (g), timing and purpose of CHO intake prior to, during and within 30-min following PA.mmol/L; b. below 3.9 mmol/L; c. below 3.0 mmol/L; d. above 10.0 mmol/L
Glucose variability 120-min before, during and 120-min after recorded structured PA sessions | 6 weeks
  Glucose variability: Standard deviation (SD) and coefficient of variance (CV) of glucose levels
Glucose variability during (at least 15-min) of habitual PA and 30-min after | 6 weeks
  Glucose variability: Standard deviation (SD) and coefficient of variance (CV) of glucose levels
Total insulin delivery 120-min before, during and 120-min after recorded structured PA sessions | 6 weeks
  Insulin delivery
Total insulin delivery during (at least 15-min) of habitual PA and 30-min after | 6 weeks
  Insulin delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — IRCM
Locations (1):
- Institut de Recherches Cliniques de Montréal (IRCM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No